CLINICAL TRIAL: NCT06355999
Title: Project 2: Levari Exp.20: 2D - Partial Feedback NOTE: Note, This is One of Many Studies Under Project 2 in the Original Grant
Brief Title: Levari Exp.20: 2D - Partial Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeremy M Wolfe, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2007p000646-F
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Form Perception; Color Perception; Decision Making
Keywords: shape perception; decision making; prevalence effects; feedback

STUDY DESIGN:
Intervention Model Description: Two groups, each receiving different feedback
Who Masked: Participant
Masking Description: Observers are naive as to the purpose of the experiment until after participation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Color Feedback (Experimental): Observers are told if the color but not if the shape was correctly identified
  Interventions: Behavioral: Color Feedback
- Shape Feedback (Experimental): Observers are told if the shape but not if the color was correctly identified
  Interventions: Behavioral: Shape Feedback

INTERVENTIONS:
Behavioral: Color Feedback — Feedback is given about the correctness of the response on the color dimension
  Arms: Color Feedback
Behavioral: Shape Feedback — Feedback is given about the correctness of the response on the shape dimension
  Arms: Shape Feedback

SUMMARY:
Suppose that observers are trying to classify a spot on the skin as normal or abnormal and suppose that the two attributes that are important are the color and shape of the spot. The investigators have found that perceptual decisions of this short are shaped by the prevalence of the target abnormality and by the feedback that observers (Os) receive. If abnormal spots are rare (low prevalence), Os will tend to become more conservative about calling spots abnormal. In this experiment, Os see items defined by color and shape. They are looking for one combination (bumpy green). Bumpy green targets can be common (50% prevalence) or rare (10%). Os in one group will get feedback about their responses based on color. The other group will receive feedback based on shape. The investigators will look for effects of prevalence and of the type of feedback. The goal is to better understand perceptual decisions in settings like clinical evaluation of skin lesions.

DETAILED DESCRIPTION:
Suppose that observers are trying to classify a spot on the skin as normal or abnormal and suppose that the two attributes that are important are the color and shape of the spot. The investigators have found that perceptual decisions of this short are shaped by the prevalence of the target abnormality and by the feedback that observers (Os) receive. If abnormal spots are rare (low prevalence), Os will tend to become more conservative about calling spots abnormal.

In this experiment, Os see items defined by color and shape. Items vary in dominant color from purple to green. Items vary in shape from relatively smooth irregular blobs (nicknamed "Bouba") to relatively bumpy blobs (nicknamed "Kiki"). Os are asked to find "Green Kikis". Since color and shape vary continuously, the border between Green Kiki and not Green Kiki will not be clear to the Os. Os will be asked to label each item as Green Kiki or not. Saying "maybe" is not an option.

The between-subject variable is the type of feedback Os receive. One set of Os will get feedback about color. That is, if the observer says "yes, this is a green kiki", they will be told only "Yes, this was a green item" or "no this was not green". The other group will get shape feedback: e.g. "Yes, this was a Kiki.".

The within-subjects variable is the target prevalence. The investigators can divide the stimuli into four quadrants: Green Kiki targets, and Green Bouba, Purple Bouba, and Purple Kiki distractors. In the high prevalence trials, 50% of the stimuli will be drawn from target quadrant (green kiki) and 17% from each of the remaining three quadrants. In the low prevalence trials, 10% of the stimuli will be drawn from the target quadrant while 30% will be drawn from each of the other three quadrants. The whole space of stimuli has 10 shape values and 10 color values for a total of 100 possible types of stimulus.

The key dependent is the proportion of target-present responses for each type of stimulus.

To analyze the data, the investigators will create a heatmap showing the percentage of times Os judge each of the 100 categories (10 colors X 10 shapes) as the target, separately for the high prevalence and low prevalence block. The investigators will calculate the response difference between the two blocks within subjects and will calculate the difference between shape and color feedback between observers.

Observers with an average accuracy below 70% will be excluded. Prior experiments have a conservative effect size of ~0.8 for differences between high and low prevalence. Some effects in experiments proposed here may have more subtle effects so power will be calculated based on an effect size of 0.6. To detect such a difference between, for instance, the 50% points on two functions like those in the data figures above, requires 26 observers to achieve alpha of 0.05 and power of 0.9. The investigators will aim for 26 observers in each condition.

ELIGIBILITY:
Inclusion Criteria:

normal color vision- 20/25 or better acuity

Exclusion Criteria:

no history of visual or oculomotor disease-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of stimuli identified as target items | Through study completion, an average one 1 year
  Participants are presented with visual stimuli from a 10 by 10 set of 100 possibilities. There are 10 levels of color (blue to green) and 10 levels of shape (smooth="Bouba" to bumpy = "Kiki", fully crossed with each other. Participants are asked to state whether an item is or is not a "green Kiki" target. For each of the 100 items, the primary outcome measure is the percentage of time that the specific item is called "Green Kiki" target.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Wolfe, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Visual Attention Lab / Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be posted on the Open Science Framework site
Supporting Information: Study Protocol, SAP, ICF
Time Frame: available after data collection, no end time
Access Criteria: openly available
URL: https://osf.io/sytaq/